CLINICAL TRIAL: NCT01323231
Title: XY-Zone Phase 1 Program Evaluation: A School-Based Dropout Prevention Program for At-Risk Male Youth
Brief Title: XY-Zone Program Evaluation: A School-Based Dropout Prevention Program for At-Risk Youth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Ronya and George Kozmetsky (RGK) Foundation (Unknown)
Responsible Party: Principal Investigator, Katherine Montgomery, PhD, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB -2010-05-0092
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Adolescent Problem Behavior at School; Risk Behavior; Truancy; Socialized
Keywords: XY-Zone; school drop-out risk; protective factors; truancy
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Communities in Schools Services (Experimental): Communities in Schools services include case management, mental health services, mentorship services, after school programs, and academic assistance.
  Interventions: Behavioral: XY-Zone

INTERVENTIONS:
Behavioral: XY-Zone — The XY-Zone works to empower students to decrease risk factors and increase protective factors through three linear treatment steps. The first step is driven by guiding principles known as the five R's: respect, responsibility, relationship, role modeling, and reaching out. Through these principles, the participant explores healthy psychosocial behaviors and thoughts in a structured 10 session group setting. The leadership step builds upon the guiding principles and employs activities exploring true leadership through 10 sessions. During the leadership step, participants organize and carry out a service learning projects in their community. The third and final step is ambassador. Those in the ambassador step become a mentor to those in step one and are "expected to explore the principles of leadership and the five R's, and determine their personal relevance to their lives as young men" (Allen, 2009, p. i).

SUMMARY:
The objective of this study is to build upon preliminary research and conduct a pilot feasibility randomized controlled trial on a promising culturally-grounded and gender-specific treatment program, the XY-Zone. The central hypothesis underlying this study purports that through receiving the XY-Zone treatment, adolescents will decrease their risk for dropping out of school. This hypothesis is supported by two years of preliminary data investigating the effectiveness of the XY-Zone.

To test the central hypothesis, the following specific aims will be pursued:

1. Identify school dropout risk and protective factors (protective factors defined as: adult support and peer support; risk factors defined as: low school attendance, inability to achieve grade promotion, substance use, delinquency, school disconnectedness, misbehavior, disconnection from healthy peers) directly changed as a result of XY-Zone intervention.
2. Determine the extent to which moderating variables (affective strength, duration in the program, family functioning, interpersonal strength, intrapersonal strength, level achieved in the program, and resiliency) effect change in outcome variables (risk and protective factors).
3. Identify participants' beliefs about the impact of the mechanisms of change (respect, responsibility, relationship, role modeling, and reaching out) on outcome variables (risk and protective factors ) to enrich understanding of quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* Students eligible to receive the XY-Zone must display one of the following risk factors:

  * academic risks (failed classes, failed state examination text, lack of class participation, and homework incompletion)
  * attendance risks (absences and tardies)
  * behavioral risks (gang involvement, substance use, classroom conduct, social skills, self-esteem, violence, delinquent conduct, and family or emotional crisis)and
  * social service issues (difficulty with the following: college readiness, life skills, health, career/employment, housing, day care, and grief or loss).

Exclusion Criteria:

* Youth who do not display any of the identified risk factors

Ages: 13 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Youth Self Report | One Year
  The Youth Self Report (Achenbach, 1991) is a 112-item scale designed for ages 11-18 years. Items are rated on a three-point scale from 0=never to 2=always true in the past 6 months. Eleven subscales can be calculated from the data, including: withdrawn, somatic complaints, anxious/depressed, social problems, thought problems, attention problems, delinquent behavior, aggressive behavior, self-destructive, and internalizing and externalizing behaviors. Scoring of subscales is gender specific. Test-retest reliability has been shown to be good (r=.84-.91).
Substance Use Self Report | One Year
  Self-report data on alcohol and other drug use will be collected through items adapted from the Adolescent DATOS survey, which was used with more than 3,000 adolescents (Kristiansen & Hubbard, 2001; Hser, Grella, et al., 2001).
School Records | One Year
  School records offer attendance, truancy, grades, grade promotion, and behavioral referral information.

SECONDARY OUTCOMES:
Behavioral and Emotional Rating Scale- II (Youth Report) | One Year
  This 57 item Likert-style scale is designed for youth ages 11-18. The BERS-II (Epstein et al., 2004) assesses six dimensions: interpersonal strength, family involvement, intrapersonal strength, school functioning, affective strength, and career and vocational strength. The BERS-II youth report has strong internal consistency (alpha=.81-.91) and good test-retest reliability (r=.84-.91).
Resilience Scale | One Year
  The resilience scale (Wagnild & Young, 1993) is a 25 item designed to measure resiliency across various populations and is appropriate for youth. Items are rated on a seven-point scale (1= strongly disagree to 7= strongly agree) and have good internal consistency (alpha= .85-.94).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Montgomery, PhD, MSSW, Principal Investigator — Washington University in Saint Louis; David W Springer, PhD, Study Chair — The University of Texas at Austin
Locations (1):
- Communities in Schools, Austin, Texas, United States

REFERENCES:
- [Background] Allen, A. (2008). The XY-Zone project evaluation of Communities in Schools-Central Texas. Independent Outcome Evaluation.
- [Background] Achenbach, T.M. (1991). Manual for the Child Behavior Checklist/ 4-18 and 1991 Profile. Burlington, VT: University of Vermont Department of Psychiatry.
- [Background] Epstein, M.H., Mooney, P., Ryser, G., & Pierce, C.D. (2004). Validity and reliability of the behavioral and emotional rating scale (2nd edition): Youth rating scale. Research on Social Work Practice, 14, 358-367.
- [Background] Hser YI, Grella CE, Hubbard RL, Hsieh SC, Fletcher BW, Brown BS, Anglin MD. An evaluation of drug treatments for adolescents in 4 US cities. Arch Gen Psychiatry. 2001 Jul;58(7):689-95. doi: 10.1001/archpsyc.58.7.689. PMID 11448377
- [Background] Kristiansen, P.L. & Hubbard, R.L. (2001). Methodological overview and research design for adolescents in the drug abuse treatment outcome studies. Journal of Adolescent Research, 16, 545-562.
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498
- [Background] Singer, J. D. and Willett, J. B. (2003). Applied longitudinal data analysis: Methods for studying change and event occurrence. New York: Oxford University Press.
- [Background] Creswell J.W. (2007). Qualitative inquiry and research design: Choosing among five approaches. 2nd ed. Thousand Oaks, CA: Sage.
- [Background] Miles M.B. & Huberman, A.M. (1994). Making good sense: Drawing and verifying conclusions. Thousand Oaks, CA: Sage.